CLINICAL TRIAL: NCT00042809
Title: Phase I Study To Determine The Safety, Tolerance And Preliminary Antineoplastic Activity Of Combined EGFR (erbB1) And HER2 (erbB2) Blockade, With OSI-774 And Trastuzumab, In Combination With Weekly Paclitaxel
Brief Title: Erlotinib, Trastuzumab, and Paclitaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02477; IDD #01-35; U01CA069853 (NIH); CDR0000069472 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Paclitaxel; Taxes; Trastuzumab; Erlotinib Hydrochloride

ARMS (1):
- Treatment (paclitaxel, trastuzumab, erlotinib hydrochloride) (Experimental): See detailed description.
  Interventions: Drug: paclitaxel; Biological: trastuzumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of combining erlotinib and trastuzumab with paclitaxel in treating patients who have advanced solid tumors. Biological therapies such as erlotinib may interfere with the growth of the tumor cells and slow the growth of the tumor. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib and trastuzumab with paclitaxel may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety, quantitative and qualitative toxic effects, maximum tolerated dose, and dose-limiting toxic effects of erlotinib when combined with paclitaxel and trastuzumab (Herceptin) in patients with advanced solid tumors.

II. Determine the relevant pharmacokinetic interactions between these agents in these patients.

III. Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, non-randomized, multicenter, dose-escalation study of erlotinib.

Intermittent schedule: Patients receive paclitaxel IV over 1 hour followed 30 minutes later by trastuzumab (Herceptin) IV over 30 minutes on days 1, 8, and 15 of each course. Patients also receive oral erlotinib once daily on days 3-28 of course 1 and on days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Continuous schedule: Once the MTD is determined using the intermittent schedule, an additional 12 patients are accrued to study the tolerability of a continuous schedule comprising paclitaxel and trastuzumab as above on days 1, 8, 15, and 22 and oral erlotinib once daily on days 3-28 during course 1 and on days 1-28 of subsequent courses using the same dose-escalation scheme as above. Courses repeat as above.

Patients are followed every 30 days.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study within 10-13.3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic solid tumor for which there are no effective standard treatment options
* HER2 positive (1+ to 3+)
* Tumor has a high likelihood of expressing epidermal growth factor receptor (EGFR)
* No evidence of leptomeningeal disease or brain metastases unless previously treated, currently asymptomatic, and off both antiepileptics and dexamethasone

  * Patients with treated brain metastases are eligible if they are without any clinical change in their brain disease status for at least 4 weeks after whole brain irradiation
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver has tumor involvement)
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* LVEF more than 50% by radionuclide ventriculogram or MUGA scan
* No significant cardiovascular disease
* No prior congestive heart failure requiring therapy
* No unstable angina pectoris
* No myocardial infarction within the past 6 months
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation

  * Patients who are unable to swallow tablets and/or who have silicon-based G-tubes may dissolve the tablets in distilled water
* No active peptic ulcer disease
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known or suspected hypersensitivity to paclitaxel
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib or other study agents
* No concurrent active infection
* No other concurrent medical condition that would preclude study participation
* No persistent grade 2 or greater neurotoxicity/neuropathy from any cause
* No psychiatric disorders or altered mental status that would preclude study participation
* No other concurrent immunotherapy
* No concurrent cytokine growth factors (e.g., colony-stimulating factors)
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy
* See Disease Characteristics
* No concurrent hormonal therapy except megestrol as an appetite stimulant or luteinizing hormone-releasing hormone agonists for prostate cancer
* See Disease Characteristics
* No concurrent radiotherapy
* No prior surgical procedures affecting absorption
* No prior EGFR-targeting therapy
* No other concurrent experimental medications or other specific antitumor therapy
* No concurrent immunosuppressant therapy
* No concurrent antiarrhythmic therapy for a ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-05; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD), graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to day 28
Response rates, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 years

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to the NCI CTC v2.0 | Up to 30 days after last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhar Beeram, Principal Investigator — Cancer Therapy and Research Center at The UT Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas, United States